CLINICAL TRIAL: NCT02949882
Title: Comparing a Probiotic and Non-probiotic Intervention in Their Ability to Improve Bowel Habits of Residents in Nursing Homes
Brief Title: Improving Bowel Habits of Elderly With Probiotics and Non-probiotics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Athena Institute, Netherlands (Other)
Collaborators: Yakult Europe BV (Industry)
Responsible Party: Principal Investigator, Eric Claassen, Prof. Dr., Athena Institute, Netherlands
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14NL-1-TLM-CON2
Record Dates: First submitted 2016-10-28; First posted 2016-10-31 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Diarrhea; Constipation
Keywords: Diarrhea; Constipation; Elderly; Nursing Homes; Probiotics; Bowel Habits
MeSH Terms: conditions — Diarrhea; Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic Intervention (Experimental): 130 Elderly participants receiving daily 65ml Yakult for 10 consecutive weeks.
  Interventions: Dietary Supplement: Yakult
- Non-Probiotic Intervention (Active Comparator): 130 Elderly participants receiving daily 65 ml of Dairy Peach Drink (AH Basic) for 10 consecutive weeks.
  Interventions: Dietary Supplement: Dairy Peach Drink (AH Basic)

INTERVENTIONS:
Dietary Supplement: Yakult — Containing at least 6,5*10^9 colony forming units (cfu) of Lactobacillus casei Shirota (LcS)
  Arms: Probiotic Intervention
Dietary Supplement: Dairy Peach Drink (AH Basic) — Commercially available dairy drink with peach flavour.
  Arms: Non-Probiotic Intervention

SUMMARY:
There is a relative high prevalence of constipation and antibiotic-associated diarrhoea (AAD) in the elderly residents of nursing homes, mainly due to high antibiotic and medication usage. Constipation and diarrhoea causes a substantial burden on lives of the frail elderly and significantly reduces the quality of life (QoL). In addition, these circumstances lead to a higher workload for healthcare workers and treatment of constipation and diarrhoea increase costs in healthcare. There are indications that the gastrointestinal microbiome is altered in conditions, such as constipation and AAD. Research indicates that probiotics show potential in the treatment of constipation, AAD and infectious diarrhoea. Probiotics can restore the aberrant gastrointestinal microbiome and thereby possibly treat/prevent constipation and diarrhoea in the frail elderly population. To illustrate, a previous pilot study of probiotic administration in elderly residents of a nursing home demonstrated a reduced prevalence of constipation and diarrhoea stool types and a higher prevalence of ideal stool types during the intervention compared to the baseline period. These promising results demand for a confirmatory study in this population.

DETAILED DESCRIPTION:
The primary objective is to assess the effect of a probiotic intervention and a non-probiotic intervention on bowel habits of elderly (>80 years on average) in several nursing homes in the Netherlands.

A randomized, double-blind, superiority, multicentre trial. In this trial a probiotic fermented milk drink will be compared to a non-probiotic drink on its potential to improve bowel habits. Both drinks are commercially available in the supermarket. After a run-in period of 2 weeks, 260 subjects will be randomized (1:1) into either the probiotic fermented milk arm (n=130) or the non-probiotic drink arm (n=130), both for a period of 10 weeks.

The study population consists of 260 frail elderly of relatively high age (>80 years old on average) living in several nursing homes in The Netherlands. One arm receives daily one bottle (65 ml) of Yakult Original (YOR), a probiotic fermented milk drink containing at least 6,5*10^9 colony forming units (cfu) of Lactobacillus casei Shirota (LcS), for 10 consecutive weeks without changing the regular diet. The other arm will receive a dairy milk drink (AH Basic Dairy Peach Drink, 65 mL) for 10 consecutive weeks, also without changing the regular diet.

The change in bowel habits of the subjects will be measured according to two main study parameters; (a) Stool-quality according to the 7-point Bristol stool chart, and (b) defecation frequency, measured as number of stools per time unit.

ELIGIBILITY:
Inclusion Criteria:

* Resident of nursing home
* Age of ≥ 70 year

Exclusion Criteria:

* Participant is seriously ill
* Immune deficient
* Intensive medication
* Life expectancy of ≤ 6 months
* Lactose intolerance
* Cow milk allergy - Stoma
* Major gastro-intestinal surgery in the past (e.g. bowel resection, gastric bypass)
* IBD
* Currently using a probiotic product, and not willing to stop this 4 weeks prior to the start of the study

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2017-04; Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Stool Quality | 10 weeks
  The primary objective is to assess the effect of a probiotic intervention and a non-probiotic intervention on bowel habits of elderly (>80 years on average) in several nursing homes in the Netherlands.
  Stool quality: will be monitored using the 7-point Bristol stool chart.
  Type 1 & 2 stools are associated with constipation, stool type 3 & 4 are characterized as ideal stools, type 5,6 & 7 stools are associated with diarrhoea.
  Bristol stool chart:
  * Type 1: Separate hard lumps, like nuts (hard to pass)
  * Type 2: Sausage-shaped, but lumpy
  * Type 3: Like a sausage but with cracks on its surface
  * Type 4: Like a sausage or snake, smooth and soft
  * Type 5: Soft blobs with clear cut edges (passed easily)
  * Type 6: Fluffy pieces with ragged edges, a mushy stool
  * Type 7: Watery, no solid pieces. Entirely liquid

SECONDARY OUTCOMES:
Defecation Frequency | 10 weeks
  Defecation frequency: will be calculated from the number of stools per time-unit.
  The frequency of defecation will be related to the Rome III criteria. For functional constipation a patient must fulfill the following diagnostic criteria:
  1. Fewer than three defecations per week
  2. Loose stools are rarely present without the use of laxatives
  3. Insuﬃcient criteria for irritable bowel syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Eric Claassen, Prof. Dr., Principal Investigator — Athena Institute, Free University of Amsterdam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Executive organisation (Clinical Research Rotterdam) — http://www.cr2o.nl